CLINICAL TRIAL: NCT07182279
Title: High Dose Rate Brachytherapy Prior to Robotic Assisted Laparoscopic Prostatectomy With Selective Adjuvant Androgen Blockade for Localized High-risk Prostate Cancer (NEOHDR-B)
Brief Title: Neoadjuvant High Dose Rate Brachytherapy Prior to Radical Prostatectomy in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Andrew Farach, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00038251
Record Dates: First submitted 2025-08-01; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: high risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decipher < 0.85 (Active Comparator): Patients will receive a single fraction of HDR-B (15Gy) 4-8 weeks prior to RALP.
  Interventions: Drug: Brachytherapy
- Decipher ≥0.85 with AAB (Active Comparator): Patients will receive a single fraction of HDR-B (15Gy) 4-8 weeks prior to RALP. In addition, patients with high genomic risk (≥0.85) will receive AAB for 12 weeks in the adjuvant setting beginning 8 weeks post RALP. Patients will receive an androgen receptor inhibitor per treating physician discretion (darolutamide 600 mg PO BID, enzalutamide 160 mg PO QD, apalutamide 240 mg PO QD, or bicalutamide 50 mg PO QD). In addition, patients will receive either a GnRH antagonist (relugolix 360 mg PO x 1 day followed by 120 mg PO QD) or a GnRH agonist (leuprolide 22.5 mg SC once or goserelin 10.8 mg SC once). Pathologically node positive patients will receive adjuvant pelvic radiation therapy as is SOC once the patient has recovered from surgery.
  Interventions: Drug: Brachytherapy

INTERVENTIONS:
Drug: Brachytherapy — All patients will receive a single fraction of HDR-B (15Gy) 4-8 weeks prior to RALP. Patients with high genomic risk or node positivity will receive short course adjuvant AAB.
  Other Names: Brachytherapy pre surgery

SUMMARY:
This is a Phase I/II trial evaluating the effectiveness of adding neoadjuvant HDR-B prior to RALP for HR-PCa patients with selective AAB for decipher high risk or pathologically node positive patients.

Patients with newly diagnosed, histologically confirmed, non-metastatic, HR-PCa who are scheduled to receive RALP will be eligible to participate in the study.

DETAILED DESCRIPTION:
Approximately, 29 cancer patients will be enrolled. Patients will receive a single fraction of HDR-B (15Gy) 4-8 weeks prior to RALP.

Patients with HR-PCa who are in the upper tercile of Decipher genomic risk (≥0.85) or have pathologically node-positive disease after lymph node dissection will receive 3 months of adjuvant AAB beginning two months post-RALP, as this is SOC for this type of patient. Node positive patients will also receive adjuvant pelvic radiation as this is SOC for this type of patient.

The primary objectives of the study will be to assess the feasibility and safety of adding HDR-B prior to RALP for patients with newly diagnosed HR-PCa and to measure per-protocol treatment compliance.

Patients will be on the study for a total of up to 27 months, including 2-3 months on active study intervention (HDR-B with RALP 4-8 weeks post HDR-B) and potentially an additional 3 months (AAB).

Study follow-ups will be performed per-protocol for up to 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have biopsy-confirmed adenocarcinoma of the prostate.
2. Subjects must have a negative bone scan and CT scan or PSMA-PET for nodal or metastatic disease.
3. Subjects must have one of the following risk factors:

   * PSA ≥20 and/or
   * Gleason score ≥8 and/or
   * Clinical or radiographic stage ≥T3a per AJCC (American Joint Committee on Cancer) 8th Edition Staging Manual and/or
   * At least two out of four of the following: PSA (Prostate Specific Antigen) 10-19.9, GS (Gleason Score) = 4+3, clinical stage = T2b/T2c, ≥50% positive biopsy cores.
4. Subjects must freely sign informed consent to enroll in the study.
5. Subjects must be medically fit to undergo surgery and HDR-B as determined by the PI.
6. Age ≥ 40
7. ECOG Performance Status (performance status is an attempt to quantify cancer patients' general well-being and activities of daily life, scores range from 0 to 5 where 0 represents perfect health and 5 represents death): 0-1.
8. No prior invasive malignancy in the past 3-years, except non-melanomatous skin cancer unless disease free for a minimum of 2 years. Carcinoma in-situ of the bladder or head and neck region is permissible.
9. Subjects must not have had prior androgen deprivation therapy in the past 6 months.

Exclusion Criteria:

1. Metastatic disease as demonstrated by bone scan, CT scan, MRI of the pelvis, or PSMA-PET.
2. Declared high-risk for anesthesia by attending cardiologist, or other physician.
3. History of prior pelvic radiation therapy.
4. Prostate gland >70 cc as assessed by MRI or TRUS.
5. Baseline IPSS >15 with medical optimization.
6. History of androgen deprivation therapy within the past 6 months (except finasteride if discontinued > 3 mo. prior to enrollment).
7. Unwilling or unable to comply with the study protocol.

   -

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 29 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to two years post RALP
  to assess the feasibility and safety of neoadjuvant HDR-B prior to RALP
Treatment Completion | up to two years post RALP
  to assess rate of treatment completion per protocol

SECONDARY OUTCOMES:
Quality of Life survey | up to two years post RALP
  to assess HRQOL as measured by International Prostate Symptom Score (IPSS) and Expanded Prostate Cancer Index Composite (Epic 26).
  These are Validated Questionnaires that will be completed by participants at Baseline and at 3, 6, 9, 12, 18, and 24 months following brachytherapy.
  The IPSS has 7 questions, and the total Score can be between 0 and 35. The IPSS has 26 questions, and the total Score can be from 0 to100.
Clinical and Pathological response | up to two years post RALP
  to asses clinical and pathological response. Clinical response will be measured with prostate specific antigen (PSA) and multi-parametric MRI of the prostate will be obtained at baseline and immediately preceding RALP (within 2 weeks).
  Pathological response will be measured with tumor assessments that will be performed at the time of prostatectomy. Margin status, treatment response (no response, partial response, complete response, extraprostatic extension, LVSI, PNI, and number of resected lymph nodes will be assessed. [ Time Frame: RALP 4-8 weeks post HDR-B]
Biochemical recurrence | up to two years post RALP
  Biochemical recurrence (BCR) will be assessed by serial serum prostate specific antigen (PSA) measurements performed at designated study visits and as clinically indicated. Two consecutive PSA measurements ≥0.2 ng/mL
Regional and distant metastasis | up to two years post RALP
  Locoregional and distant metastasis-free survival will be assessed by scheduled and symptom-driven imaging (CT, MRI, bone scan, or PET per protocol) and biopsy when clinically indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Farach, MD, Principal Investigator — The Methodist Hospital Reseach Institute
Locations (1):
- Houston Methodist, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No